CLINICAL TRIAL: NCT04943484
Title: [The iGreenGO Study]. Investigation About the Clinical Value of Indocyanine Green Imaging Fluorescence (NIR/ICG) Technology as a Modifier of Surgeon's Conduct During Curative Treatment of Advanced Gastric Cancer. Study Protocol for a Western, Observational, Prospective, Multicentric Study
Brief Title: ICG (Indocyanine Green) Imaging Fluorescence Technology in Surgical Treatment of Advanced Gastric Cancer
Acronym: iGreenGO
Status: Recruiting | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 380-09062021
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer
Keywords: advanced; gastric cancer; indocyanine green; ICG; surgery; D2 lymphadenectomy; surgical conduct
MeSH Terms: conditions — Stomach Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastric cancer: Male and female subjects, over 18 years of age, with histological diagnosis of locally advanced gastric carcinoma (AGC), surgically resectable, without evidence of distant metastases (cT2-T4a; N0-3; M0) for which a surgical intervention with curative purposes is indicated both as a first treatment and following preoperative neoadjuvant chemotherapy
  Interventions: Procedure: imaging fluorescence NIR/ICG

INTERVENTIONS:
Procedure: imaging fluorescence NIR/ICG — Preoperative upper GI endoscopy (UGE) UGE with submucosal injection of 2ml of ICG 0.125mg/ml solution to four peritumoral sites 15-20 hours before surgery Surgery D2 Distal gastrectomy with dissection of 1, 3, 4sb, 4sd, 5, 6, 7, 8a, 9, 11p, 12a lymph node stations (LNS) D2 Total gastrectomy with dissection of 1, 2, 3, 4sa, 4sb, 4d, 5, 6, 7, 8a, 9, 11p, 11d, 12a LNS Intraoperative NIR/ICG technology, "change of surgical conduct" (CSC) A visualization of the operative field (OF) with NIR/ICG technology is performed at the beginning of surgery and before to dissect each LNS. Subsequently, surgery is performed "with the naked eye".
  At the end, a visualization of the OF is performed using NIR/ICG technology to verify whether residual lymph nodes in each D2 nodal station exist. CSC is defined as the occurring of the following situation: in case of persistence of nodal fluorescence in D2 nodal stations, the completion of the dissection of the residual nodal fluorescent structures.
  Other Names: indocyanine green

SUMMARY:
The iGreenGO Study aims to investigate whether the intraoperative application of NIR/ICG technology is associated with a change in the surgical conduct (CSC) during curative-intent gastrectomy with D2 lymphadenectomy in a cohort of Western patients affected by AGC. The preoperative clinical variables potentially associated with CSC will be also investigated

DETAILED DESCRIPTION:
Near infra-red/ indocyanine green imaging fluorescence (NIR/ICG) technology is showing promising results in several fields of surgical oncology.

The clinical value of NIR/ICG (near infrared range/indocyanine green) technology in surgical treatment of advanced gastric cancer (AGC) is not clearly established and data regarding whether its application is associated with a change of the intraoperative surgical conduct are lacking in literature.

This is the "iGreenGO (indocyanine Green Gastric Observation) Study" protocol: an international, prospective, multicentre, study.

Study population will be a cohort of western patients who will undergo preoperative upper gastrointestinal endoscopy at the most 20 hours before surgery (intraoperative endoscopic injection before starting surgical dissection is also allowed) with submucosal peritumoral ICG injection and curative-intent gastrectomy with D2 lymphadenectomy for locally AGC.

The primary endpoint will be the incidence of "change of the surgical conduct" (CSC) at the moment of intraoperative NIR/ICG technology activation after a D2 lymphadenectomy performed "with the naked eye". Secondary endpoints will be the preoperative clinical variables potentially associated with CSC, the pattern of abdominal fluorescence distribution according to tumor and patient characteristics, the number of additional lymph nodes retrieved using NIR/ICG technology, the incidence of stage migration due to NIR/ICG application, 90-day morbidity and mortality The iGreenGO Study will be the first Western study to investigate the clinical role of NIR/ICG technology for surgical treatment of AGC in a large cohort of western patients. Results from the present study could provide novel information about which help NIR/ICG technology can supply to surgeons during lymphadenectomy for AGC and the patterns of ICG abdominal fluorescence distribution according to tumor and patient characteristics, which are unanswered questions at present time.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years old
* Preoperative histologically proven adenocarcinoma of the upper, middle or lower part of the stomach.
* Advanced disease (Staged cT2-T4a, N0-3;M0 according to 8th edition of the AJCC TNM Staging System) at diagnosis, in which resection can be safely achieved by distal or total gastrectomy with D2 lymphadenectomy via a minimally invasive (laparoscopic or robotic) approach, either as first treatment or after neoadjuvant treatment
* No distant metastasis, no direct invasion of pancreas, spleen or other organs nearby in the preoperative and intraoperative examinations
* Written informed consent

Exclusion criteria

* Women during pregnancy or breast-feeding
* History of previous upper abdominal surgery (laparoscopic cholecystectomy will be allowed)
* History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
* History of allergy to iodine agents
* Cancer located at the esophago-gastric junction (Siewert I, II, III tumors 29)
* Patients candidates to transthoracic esophagectomy, transhiatal extended gastrectomy or proximal gastrectomy
* History of previous neoadjuvant chemotherapy (except perioperative chemotherapy for gastric cancer) or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects, over 18 years of age, with histological diagnosis of locally advanced gastric carcinoma (AGC), surgically resectable, without evidence of distant metastases (cT2-T4a; N0-3; M0) for which a surgical intervention with curative purposes is indicated both as a first treatment and following preoperative neoadjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Surgical conduct | During surgical intervention (hours)
  Incidence of "change of the surgical conduct" (CSC) at the moment of intraoperative NIR/ICG technology activation after a D2 lymphadenectomy performed "with the naked eye"

SECONDARY OUTCOMES:
Nodal fluorescence distribution | During surgical intervention (hours)
  Pattern of nodal fluorescence distribution according to tumor and patient characteristics
Clinical variables associated with change of the surgical conduct | During surgical intervention (hours)
  Identification of preoperative clinical variables potentially associated with change of the surgical conduct

CONTACTS AND LOCATIONS:
Overall Officials: Pietro M Lombardi, MD, Principal Investigator — Division of Minimally Invasive Surgical Oncology, Niguarda Cancer Center, ASST Grande Ospedale Metropolitano Niguarda
Locations (1):
- ASST GOM Niguarda, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Monthly planned meeting among researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 4 years
Access Criteria: Participant centres